CLINICAL TRIAL: NCT06211725
Title: The VANGAS-Trial. The Value of Neurofilament Light Chain and Glial Fibrillary Acid Protein in the Blood of Patients With Asymptomatic Carotid Artery Stenosis
Acronym: VANGAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: VANGAS
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Stenosis Asymptomatic; Carotid Artery Diseases; Carotid Artery Plaque
Keywords: Carotid Artery Stenosis; Carotid Artery Plaque; Carotid Artery Disease; Carotid Artery Stenosis asymptomatic; Carotid artery stenosis biomarker; carotid artery nfl; carotid artery gfap; Carotid Artery Plaque Biomarker
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neurovascular patients

SUMMARY:
Stroke is the second leading cause of death and the third leading cause of disability worldwide. The cause is usually either a blockage or a severe narrowing of a cerebral artery. An important part of stroke prevention is the diagnosis and clarification of stenosis in the arteries supplying the brain, both inside and outside the skull, in order to diagnose a high-grade stenosis at an early stage and offer the patient revascularization. In particular, asymptomatic carotid artery stenosis confronts the diagnosing physician with the question of whether revascularisation is necessary.

Risk factors for stroke in asymptomatic carotid artery stenosis include contralateral TIA or cerebral infarction, male gender, rapid progression of the degree of stenosis, plaque morphology, clinically silent cerebral infarctions, Doppler sonographic evidence of microemboli or reduced vasomotor reserve. An established biomarker does not exist at this time. A candidate for such a biomarker in the blood is the protein "neurofilament light chain" (NFL), which is already established in the diagnosis of dementia. As a component of the cytoskeleton of neurons, it is released into the patient's blood when the cells are damaged and can be measured there. Another candidate is glial fibrillary acid protein (GFAP), a part of the cytoskeleton of glial cells that is also released into the blood when glial cells are damaged. A systematic investigation of the value of neurofilament light chain and the glial fibrillary acidic protein in the blood of patients with asymptomatic carotid stenosis is still lacking. VANGAS determines the value of NFL and GFAP from the blood of patients with asymptomatic carotid stenosis to determine associations with the degree of stenosis, the natural course of the stenosis (increase or decrease) and possible symptoms of the stenosis as well as the functional outcome after symptomatic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 60- 80 years
* 0-100 % stenosis of the internal carotid artery

Exclusion Criteria:

* Neurodegenerative diseases such as any form of dementia or Parkinson's disease
* Polyneuropathy
* Multiple sclerosis
* Stroke (ischaemic or haemorrhagic) within the last 12 months
* Transient ischaemic attack within the last 12 months
* Neurotrauma within the last 12 months
* Atrial fibrillation

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are included from our and the cooperating neurological clinics and practices
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of NF-L/GFAP with degree of stenosis (NASCET-Criteria) | 24 months
  The amount of NF-L and GFAP in the blood of patients with stenosis of a brain-supplying artery correlates with the degree of the stenosis.

SECONDARY OUTCOMES:
Correlation of NF-L/GFAP with functional outcome (modified rankin scale) | 24 months
  The amount of NF-L and GFAP in the blood of patients with stenosis of a brain-supplying artery correlates with functional outcome after symptomatic stenosis
Correlation of NF-L/GFAP with progression of stenosis (NASCET-Criteria) | 24 months
  The amount of NF-L and GFAP in the blood of patients with stenosis of a brain-supplying artery correlates with the progression of the stenosis (increase or decrease).
Correlation of NF-L/GFAP with future cerebral ischemia (Stroke / TIA) | 24 months
  The amount of NF-L and GFAP in the blood of patients with stenosis of a brain-supplying artery allows differentiation between future symptomatic and asymptomatic stenosis

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided